CLINICAL TRIAL: NCT05815524
Title: Physical Activity in Patients With Parkinson's Disease: a "Disease Modifying" Intervention?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Overlapping studies
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 4938
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): physical activity protocol
  Interventions: Other: Physical activity training

INTERVENTIONS:
Other: Physical activity training — training on treadmill

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disease characterized by bradykinesia, rigors, and tremor at rest. Distinctive neuropathological signs include progressive loss of dopaminergic neurons in the Substantia nigra pars compacta (SNpc) and the presence of immunoreactive protein inclusions for α-syn, Lewy bodies (LB). The clinical phenotype is heterogeneous, both from a motor and non-motor point of view. Furthermore, the prognosis and response to drugs are highly variable and poorly predictable. To date, there are no biomarkers capable of early identification of clinical phenotypes and of predicting response to therapy. This constitutes a serious limit that probably represents one of the causes of the failure of the experimentation of the disease modifying therapies tested up to now (for example the anti-α-sin antibodies). Certainly, a deeper understanding of disease pathogenesis is needed to address these unsolved problems.

Oxidative stress and inflammation have critical roles in PD, especially in the prodromal and early stages of PD, as they contribute to pathological progression and also trigger potentially devastating neuroprotective responses, especially in the early stages. Consequently, soluble mediators of these processes may represent potential markers of prodromal phases of the disease.

Inflammation is a key factor in the initiation and propagation of a-syn aggregates and the contribution of microglial activation to a-syn pathology has been highlighted recently. Elevated a-syn specific T cell responses may be present years before the diagnosis of motor PD, suggesting a role of neuroinflammation in PD pathogenesis and early diagnosis. Furthermore, studies in rats overexpressing a-syn support the idea that reducing neuroinflammation could improve symptoms in early Parkinson's disease. In particular, drug-targeted anti-inflammatory approaches in a-syn rats prevent central and peripheral inflammation, as well as neuronal dysfunction and motor motor impairment.

It is also increasingly evident that panels that combine different biomarkers, with a multimodal approach, are more sensitive and specific, better reflecting the complexity of pathophysiological mechanisms. In fact, the diagnostic sensitivity of some CSF biomarker panels of neurodegeneration in distinguishing between atypical parkinsonisms and Parkinson's disease has been demonstrated. These markers, as well as in the cerebrospinal fluid, can be measured in the serum, albeit with reduced specificity, and in exosomes of central origin, which have recently been described and analyzed also in cohorts of patients with Parkinson's disease.

In addition to pharmacological approaches, attention has recently been paid to non-pharmacological therapeutic approaches, such as physical activity.

In particular, studies on PD patients show that aerobic exercise improves motor performance by increasing BDNF levels and reducing inflammation. Retrospective studies have found that moderate to vigorous exercise in midlife may protect against PD. In 2018, a phase 2 study investigated the response to treadmill exercise performed at two different intensities (high and moderate) by de novo PD patients, reporting a beneficial effect of moderate treadmill exercise. Although aerobic exercise appears to be the most effective, several studies have used a variety of exercise programs to demonstrate options available for those who cannot physically perform aerobic exercise. In PD patients, physical activity also appears to have beneficial effects on cognition, mood, and sleep quality. Preclinical findings support the hypothesis that physical activity exerts its beneficial effect by increasing levels of BDNF and anti-inflammatory cytokines and inhibiting pro-inflammatory factors.

In this study the investigators will measure changes in clinical scales and biomarkers in patients who undergo either an intensive physical activity protocol or continue their routine sedentary life.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD defined according to MDS criteria
* Hoehn & Yahr Stage 1-3
* Stable dopaminergic therapy in the previous month
* Duration of disease of at least 3 years
* MMSE > 24/30
* Age between 45-70 years
* Signature of the informed consent to participate in the study in question

Exclusion Criteria:

* Contraindications to the practice of physical activity as required by the European Society of Cardiology 2020 guidelines
* Practice of regular sporting activity for more than 150 minutes per week
* Serious orthopedic pathologies
* Severe psychiatric disorders
* Inflammatory or autoimmune diseases
* Active oncological pathologies
* Known cardiovascular and/or cardiorespiratory pathologies that may contraindicate or influence the performance of the motor program (ischaemic heart disease, arterial hypertension not under pharmacological treatment, primary or secondary non-Parkinson-related cardiomyopathies and/or valve diseases, channelopathies, anemia, heart failure, COPD pulmonary hypertension, bronchial asthma).

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
clinical response | 2 years
  To measure motor performance in a population of PD patients before and after a physical activity protocol, compared to a sedentary population using the Unified Parkinson's disease rating scale (UPDRS) (min 0- max 260, better clinical conditions has lower scores)

SECONDARY OUTCOMES:
biomarkers | 2 years
  To measure peripheral biomarkers of neurodegeneration, neurotrophic and inflammation in a population of PD patients before and after a physical activity protocol, compared to a sedentary population.
  Biomarkers related to axonal damage (total tau (t-Tau), neurofilament light chain, (NfL), and phosphorylated neurofilament heavy chain, (p-NfH), synaptic dysfunction (a-synuclein (a-syn) and neurogranin, (Ng)), neuroinflammation (soluble triggering receptor expressed on myeloid cells 2, sTREM2, and chitinase-3- like protein 1, YKL-40, IL1b, IL4, IL5, IL6, IL10, IL17, IFNg, TNF) will be analysed in blood (for all the biomarkers, ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rita Bentivoglio, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Flavia Torlizzi, Roma, Italy